CLINICAL TRIAL: NCT05957445
Title: Personalized Brain Functional Sector-guided Multi-target Continuous Theta Burst Stimulation Therapy for Aphasia After Stroke: a RCT
Brief Title: pBFS-guided Multi-target cTBS for Aphasia After Stroke
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Changping Laboratory (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CPSA06HB60
Record Dates: First submitted 2023-07-14; First posted 2023-07-24 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2024-07

CONDITIONS: Stroke; Aphasia
MeSH Terms: conditions — Stroke; Aphasia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- active cTBS group (Active Comparator): active cTBS combined with speech language therapy
  Interventions: Device: active continuous Theta Burst Stimulation
- sham cTBS group (Sham Comparator): sham cTBS combined with speech language therapy
  Interventions: Device: sham continuous Theta Burst Stimulation

INTERVENTIONS:
Device: active continuous Theta Burst Stimulation — Each patient will receive a series of stimulation sequences, including a 600-pulse cTBS targeting at the right IFG, followed by a 600-pulse cTBS targeting at the right STG, and subsequently a 600-pulse cTBS targeting at the right SFG. This sequence will be repeated once more (a total of 3600 pulses daily). Each patient will receive a 3-week treatment period, consisting of 5 consecutive workdays each week.
  Arms: active cTBS group
Device: sham continuous Theta Burst Stimulation — Each patient will receive a series of stimulation sequences，including a 600-pulse sham cTBS targeting at the right IFG, followed by a 600-pulse sham cTBS targeting at the right STG, and subsequently a 600-pulse sham cTBS targeting at the right SFG. This sequence will be repeated once more (a total of 3600 pulses daily). Each patient will receive a 3-week treatment period, consisting of 5 consecutive workdays each week.
  Arms: sham cTBS group

SUMMARY:
In this study, a randomized, double-blind, parallel-controlled trial was employed to evaluate the effectiveness and safety of personalized brain functional sectors (pBFS) technology-guided continuous theta burst stimulation (cTBS) on the inferior frontal gyrus (IFG) combined with the superior temporal gyrus (STG) and the superior frontal gyrus (SFG) for language function recovery in post-stroke aphasic patients.

DETAILED DESCRIPTION:
Increasing evidence suggests that rTMS has been effective in treating various psychological and neurological diseases, including treating post-stroke symptoms. Using the personalized brain functional sectors (pBFS) technique, investigators could precisely identify individualized brain functional networks and the personalized language-related stimulation site based on the resting-state functional MRI data. The current study proposes to conduct a double-blinded, randomized and parallel controlled design trial, to investigate the efficacy and safety of pBFS-guided multi-target rTMS intervention in post-stroke aphasic patients.

Subjects will be randomly assigned to the following two groups: active continuous TBS (cTBS) group, or a sham control group. The allocation ratio will be 1:1. The stimulation protocol consisted of a 3-week treatment, with 5 consecutive workdays each week (totally 15 day-treatment). The stimulation procedure will be assisted with real-time neuronavigation to ensure its precision.

ELIGIBILITY:
Inclusion Criteria:

* The patient's age ranges from 35 to 75 years old (including 35 and 75 years old);
* Meet the diagnostic criteria for ischemic stroke (according to the guidelines developed by the American Heart Association/American Stroke Association in 2019 and the guidelines developed by the Neurology Branch of the Chinese Medical Association in 2018) or meet the diagnostic criteria for hemorrhagic stroke (according to the guidelines developed by the American Heart Association/American Stroke Association in 2022 and the guidelines developed by the Neurology Branch of the Chinese Medical Association in 2019) ，with lesions located in the left hemisphere, and a duration of illness ranging from 15 days to 6 months.
* Diagnosed as aphasia patient according to the Chinese version of Western Aphasia Battery (WAB), with a WAB-aphasia quotient of less than 93.8 points;
* First onset of stroke;
* Normal language function before the onset of stroke, and the patient's native language is Chinese with at least 6 years of education;
* Understand the trial and signed the informed consent form.

Exclusion Criteria:

* Combined dysarthria (NIHSS item 10 score ≥2 points);
* Aphasia caused by bilateral hemisphere stroke, brain tumor, traumatic brain injury, Parkinson's disease, motor neuron disease, or other diseases；
* Patients with implanted electronic devices such as cardiac pacemakers, cochlear implants, or other metal foreign bodies, or those with MRI contraindications such as claustrophobia or TMS treatment contraindications;
* History of epilepsy;
* Patient with concomitant severe systemic diseases affecting the heart, lungs, liver, kidneys, etc., and uncontrolled by conventional medication, as detected and confirmed through laboratory testing and examination;
* Patients with consciousness disorders (NIHSS 1(a) score ≥1);
* Patients with malignant hypertension;
* Patients with severe organic diseases, such as malignant tumors, with an expected survival time of less than 1 year;
* Patients with severe hearing, visual, cognitive impairment or inability to cooperate with the trial;
* Patients with severe depression, anxiety, or diagnosed with other mental illnesses that prevent them from completing the trial;
* Patients who have received other neuromodulation treatments such as TMS, transcranial electric stimulation, etc. in the 3 months prior to enrollment;
* Patients with a history of alcoholism, drug abuse, or other substance abuse;
* Patients with other abnormal findings that the researchers judge are not suitable for participation in this trial;
* Patients who are unable to complete follow-up due to geographical or other reasons;
* Women of childbearing age who are currently pregnant, breastfeeding, or planning or may become pregnant during the trial;
* Patients who are currently participating in other clinical trials.

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-08-23 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Change in the Western Aphasia Battery scores | baseline, end of the 3-week therapy
  The first four subsets of the WAB (Spontaneous Speech, Auditory verbal comprehension, Repetition, Naming and word finding) will be used to evaluate the participants' language ability impairments. A Chinese adapted version of WAB will be used. The scores from all four subsets will be calculated as an Aphasia Quotient (ranging from 0 to 100), with lower Aphasia Quotients indicating poorer language abilities.

SECONDARY OUTCOMES:
Change in the Western Aphasia Battery scores | baseline, end of the 5-day therapy, 90 days after treatment initiation
  The first four subsets of the WAB (Spontaneous Speech, Auditory verbal comprehension, Repetition, Naming and word finding) will be used to evaluate the participants' language ability impairments. A Chinese adapted version of WAB will be used. The scores from all four subsets will be calculated as an Aphasia Quotient (ranging from 0 to 100), with lower Aphasia Quotients indicating poorer language abilities.
Boston Diagnostic Aphasia Examination Severity Ratings | baseline, end of the 3-week therapy，90 days after treatment initiation
  The Boston Diagnostic Aphasia Examination (BDAE) Severity Ratings is a clinical tool used to evaluate the severity and type of aphasia in individuals. The assessment includes four domains: communication abilities, language content, speech sound production and response abilities.BDAE severity ratings range from level 0 to level 5, with lower scores indicating more severe aphasia.
Token test | baseline，end of the 3-week therapy，90 days after treatment initiation
  The Token Test is a language assessment tool used to evaluate a person's ability to understand spoken language and follow instructions. Each correct response in each task is awarded one point, typically. Different point values may be assigned based on the complexity of the task. The total score is calculated by adding up the accumulated scores across all tasks. The total scores range from 0 to 36, with higher scores indicating better language abilities.
Chinese-version Stroke and Aphasia Quality of Life Scale 39-generic version (SAQOL-39g) | baseline，end of the 3-week therapy，90 days after treatment initiation
  The SAQOL-39g is a quality of life assessment tool that is used to evaluate the impact of stroke and aphasia on a patient's quality of life. It consists of 39 items that cover a range of domains related to the patient's quality of life, such as communication, physical functioning, mood, and social support. The items are rated on a 5-point Likert scale ranging from "not at all" to "very much", with higher scores indicating better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Hesheng Liu, PhD, Study Chair — Changping Laboratory
Locations (3):
- China (3):
  - Affiliated Hospital of Hebei University, Baoding, Hebei
  - Affiliated Hospital of Chengde Medical University, Chengde, Hebei
  - Hebei General Hospital, Shijiazhuang, Hebei

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Huang J, Ren J, Xie W, Pan R, Xu N, Liu H. Personalised functional imaging-guided multitarget continuous theta burst stimulation for post-stroke aphasia: study protocol for a randomised controlled trial. BMJ Open. 2024 May 15;14(5):e081847. doi: 10.1136/bmjopen-2023-081847. PMID 38754874